Athens, 1.11.2025

## **Unique Protocol ID: RAKITZI CYSTIC FIBROSIS**

Official title of the study: The effectiveness and efficacy of an online group cognitive behavioral psychotherapy in patients with cystic fibrosis and caregivers in comparison to control groups by the Hellenic Cystic Fibrosis Association A Randomized Controlled Trial

Brief title: The effectiveness and efficacy of an online cognitive behavioral psychotherapeutic program (RAKITZIHCFA)

NCT: not available

Sponsor: Dr. Stavroula Rakitzi

Dr. phil., Dipl.-Psych., Stavroula Rakitzi

Clinical psychologist and cognitive behavioral psychotherapist

Private practice

ILISION 34 15771 Athens Greece

2111180571

6989766935

Stavroula@Rakitzi.onmicrosoft.com

srakitzi@gmail.com

Description linkedin Stavroula Rakitzi

ORCID: http://0000-0002-5231-6619

In collaboration with the Hellenic Cystic Fibrosis Association

(www.cysticfibrosis.gr/en)

President: Anna Spinou

Karaiskaki street 28 105 54 Athens Greece

Tel: +302110137700, +306944255853

E-mail: info@cysticfibrosis.gr

## Informed consent to the research protocol

Dr. Stavroula Rakitzi, a clinical psychologist and cognitive behavioral psychotherapist will conduct a research protocol in collaboration with the Hellenic Cystic Fibrosis Association in Athens Greece regarding the effectiveness and efficacy of an online group cognitive behavioral psychotherapy for patients with cystic fibrosis and for caregivers in comparison with control groups. Participation in the therapy group or the control group is the result of a draw because this study is a randomized control trial.

The research protocol begins on 15 11.2025. The tests will be administered before the therapy, after the therapy and in a follow-up after 6 months (24 weeks). The research protocol will be registered at ClinicalTrials.gov.

The test results will be used for statistical analysis to research the effectiveness and efficacy of the treatment. Results will be anonymous, and no personal data will be displayed from any individual participating in the groups. I will let you know about the results. The results will be published in a scientific journal or a book. My participation in this research protocol is voluntary. I certify that I have been informed of the above and that I agree with them.

| Name | Signature |
|------|-----------|
| | Name |